CLINICAL TRIAL: NCT03370692
Title: Development and Validation of a Prognostic Score in the Very Old ICU Patients (≥80 Years)
Brief Title: Prognostic Score in the Very Old ICU Patients
Acronym: VIP2
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Helse Vest (Other); European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Hans Flaatten, Professor, University of Bergen
Other Study IDs: VIP2
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Aged, 80 and Over; Critical Care
Keywords: Outcome; Survival; Prognostication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cognitive assesment, Frailty assessment — Asking relatives (using a structured questionaire) about cognitive function at admission , likewise about frailty using the Clinical Frailty Score

SUMMARY:
The two main aims of the study:

1. To investigate the relation of Frailty, Activity of daily life (ADL), Cognitive functions and Co-morbidity on survival at 30 days (and 6 months in a substudy)
2. From the results design a prognostic score that will be validated using a subpopulation of the study cohort

Two secondary aims a

1. Survival at 6 months (in a subpopulation of the study)
2. An inter-rater validation of the Clinical Frailty Score (CFS) (in a subpopulation)

Substudies are planned with regards to the different admission categories, in particular:

* trauma
* acute respiratory failure
* sepsis
* combined respiratory and circulatory failure
* medical neurological conditions In some of the substudies similar groups from the VIP1 study that uses the same admission categories (except planned admissions) will be merged.

DETAILED DESCRIPTION:
Frailty to be registered by the Clinical Frailty Scale (CFS), 1-9 point Activity of Daily life (ADL) with Katz ADL form: 0-6 points Cognition to be described by Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) questionaire, 16 questions to be asked the care-givers Co-morbidity by listing the major comorbidity with Yes or No (Yes= 1 point) and with the number of regular drugs prescribed

ELIGIBILITY:
Inclusion Criteria:

* ≥80 admitted to an ICU as an emergency case

Exclusion Criteria:

* elective admissions

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Critical ill patients admitted to the ICU ≥ 80 years
Sampling Method: Non-Probability Sample
Enrollment: 3900 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
30 days survival | 30 days
  Proportion alive after 30 days

SECONDARY OUTCOMES:
Developement of a prognostic score | 6 months
  Developement and subsequent validation of a prognostic score from data revealed in the study: Frailty, Comorbidity, Activity of Daily life and Cognition. This score is non-existent at the moment, it is a score we will develope and test within the cohort-. No further description can be given before study is finished and analysed.
6 months survival | 6 months
  Proportion alive after 6 months
Inter-rater validation of Clinical Frailty Scale (CFS) | At admission
  The CFS is a simple visual scale of frailty from 1 to 9 (increasing frailty). We will in a subset of our patients use two raters to perform frailty score and compare their results using inter-rater variability tests.

OTHER OUTCOMES:
Survival analysis in pre-defined subgroups: Admission categories, use of therapeutic procedures, end-of-life desicion | Up to 6 months
  Proportions alive after 30 days and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Lange DW, Soliman IW, Leaver S, Boumendil A, Haas LEM, Watson X, Boulanger C, Szczeklik W, Artigas A, Morandi A, Andersen F, Jung C, Moreno R, Walther S, Oeyen S, Schefold JC, Cecconi M, Marsh B, Joannidis M, Nalapko Y, Elhadi M, Fjolner J, Guidet B, Flaatten H; VIP2 study group. The association of premorbid conditions with 6-month mortality in acutely admitted ICU patients over 80 years. Ann Intensive Care. 2024 Mar 30;14(1):46. doi: 10.1186/s13613-024-01246-w. PMID 38555336
- [Derived] Mousai O, Tafoureau L, Yovell T, Flaatten H, Guidet B, Beil M, de Lange D, Leaver S, Szczeklik W, Fjolner J, Nachshon A, van Heerden PV, Joskowicz L, Jung C, Hyams G, Sviri S. The role of clinical phenotypes in decisions to limit life-sustaining treatment for very old patients in the ICU. Ann Intensive Care. 2023 May 10;13(1):40. doi: 10.1186/s13613-023-01136-7. PMID 37162595
- [Derived] Beil M, van Heerden PV, de Lange DW, Szczeklik W, Leaver S, Guidet B, Flaatten H, Jung C, Sviri S, Joskowicz L. Contribution of information about acute and geriatric characteristics to decisions about life-sustaining treatment for old patients in intensive care. BMC Med Inform Decis Mak. 2023 Jan 6;23(1):1. doi: 10.1186/s12911-022-02094-z. PMID 36609257
- [Derived] Guidet B, Jung C, Flaatten H, Fjolner J, Artigas A, Pinto BB, Schefold JC, Beil M, Sigal S, van Heerden PV, Szczeklik W, Joannidis M, Oeyen S, Kondili E, Marsh B, Andersen FH, Moreno R, Cecconi M, Leaver S, De Lange DW, Boumendil A; VIP2 and COVIP study groups. Increased 30-day mortality in very old ICU patients with COVID-19 compared to patients with respiratory failure without COVID-19. Intensive Care Med. 2022 Apr;48(4):435-447. doi: 10.1007/s00134-022-06642-z. Epub 2022 Feb 26. PMID 35218366
- [Derived] Bruno RR, Wernly B, Kelm M, Boumendil A, Morandi A, Andersen FH, Artigas A, Finazzi S, Cecconi M, Christensen S, Faraldi L, Lichtenauer M, Muessig JM, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Valentin A, Watson X, Leaver S, Boulanger C, Walther S, Schefold JC, Joannidis M, Nalapko Y, Elhadi M, Fjolner J, Zafeiridis T, De Lange DW, Guidet B, Flaatten H, Jung C; VIP2 study group. Management and outcomes in critically ill nonagenarian versus octogenarian patients. BMC Geriatr. 2021 Oct 19;21(1):576. doi: 10.1186/s12877-021-02476-4. PMID 34666709
- [Derived] Fronczek J, Polok K, de Lange DW, Jung C, Beil M, Rhodes A, Fjolner J, Gorka J, Andersen FH, Artigas A, Cecconi M, Christensen S, Joannidis M, Leaver S, Marsh B, Morandi A, Moreno R, Oeyen S, Agvald-Ohman C, Bollen Pinto B, Schefold JC, Valentin A, Walther S, Watson X, Zafeiridis T, Sviri S, van Heerden PV, Flaatten H, Guidet B, Szczeklik W; VIP1; VIP2 study group. Relationship between the Clinical Frailty Scale and short-term mortality in patients >/= 80 years old acutely admitted to the ICU: a prospective cohort study. Crit Care. 2021 Jul 1;25(1):231. doi: 10.1186/s13054-021-03632-3. PMID 34210358
- [Derived] Wernly B, Beil M, Bruno RR, Binnebossel S, Kelm M, Sigal S, van Heerden PV, Boumendil A, Artigas A, Cecconi M, Marsh B, Moreno R, Oeyen S, Bollen Pinto B, Szczeklik W, Leaver S, Walther SM, Schefold JC, Joannidis M, Fjolner J, Zafeiridis T, de Lange D, Guidet B, Flaatten H, Jung C; VIP2 study group. Provision of critical care for the elderly in Europe: a retrospective comparison of national healthcare frameworks in intensive care units. BMJ Open. 2021 Jun 3;11(6):e046909. doi: 10.1136/bmjopen-2020-046909. PMID 34083342
- [Derived] Wernly B, Bruno RR, Kelm M, Boumendil A, Morandi A, Andersen FH, Artigas A, Finazzi S, Cecconi M, Christensen S, Faraldi L, Lichtenauer M, Muessig JM, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Niederseer D, Valentin A, Watson X, Leaver S, Boulanger C, Walther S, Schefold JC, Joannidis M, Nalapko Y, Elhadi M, Fjolner J, Zafeiridis T, De Lange DW, Guidet B, Flaatten H, Jung C. Sex-specific outcome disparities in very old patients admitted to intensive care medicine: a propensity matched analysis. Sci Rep. 2020 Oct 29;10(1):18671. doi: 10.1038/s41598-020-74910-3. PMID 33122713